CLINICAL TRIAL: NCT00409396
Title: Urinary PGE-M, A Metabolite of PGE2: A Novel Biomarker of Ulcerative Colitis Disease
Brief Title: A Study to Determine Whether Urinary PGE-M Levels Correlate With Ulcerative Colitis Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, David Schwartz, Principal Investigator, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Urinary PGE-M UC
Record Dates: First submitted 2006-12-05; First posted 2006-12-08 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2014-11

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative; Colitis; PGE-M; fecal calprotectin; disease biomarkers
MeSH Terms: conditions — Colitis, Ulcerative; Ulcer; Colitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Fecal calprotectin and urinary PGEm levels will be tested on all participants.
  Interventions: Procedure: Urinary PGEm level; Procedure: fecal calprotectin

INTERVENTIONS:
Procedure: Urinary PGEm level — Level of PGEm in urine compared to CRP and fecal calprotectin levels in patients with ulcerative colitis.
Procedure: fecal calprotectin — Level of fecal calprotectin in comparison to urinary PGEm and serum CRP levels.

SUMMARY:
The purpose of this study is to determine whether urinary PGE-M levels correlate with Ulcerative Colitis Disease activity and to compare how well urinary PGEm correlates with other noninvasive biomarkers of disease activity such as CRP and fecal calprotectin.

DETAILED DESCRIPTION:
The available clinical measures of ulcerative colitis activity can be overly influenced by functional symptoms. Placebo response rates in clinical trials are high. Several non-invasive biomarkers are currently available for assessing IBD disease activity including erythrocyte sedimentation rate, c-reactive protein and fecal calprotectin. Although these markers hold some promise, their performance is less than ideal. what is needed is a simple, non-invasive biologic measure of UC disease.

Cyclooxygenase-2 (COX-2) is involved in prostaglandin E2 (PGE2) synthesis and is expressed in epithelial inflammatory conditions and some cancers. We have developed an assay to quantify the major urinary metabolite of PGE2, PGE-M. PGE-M has been previously shown to be elevated in the urine of patients with advanced colorectal neoplasia relative to controls. We recently showed that PGEm was a sensitive and specific marker of Crohn's disease activity (Accepted for publication at DDW 2006).

ELIGIBILITY:
Inclusion Criteria:

* Outpatient male or female 18 years or older
* Confirmed diagnosis of ulcerative colitis
* Informed consent obtained
* Able to give blood, urine and stool samples
* Will undergo a diagnostic colonoscopy of part of routine Ulcerative Colitis care

Exclusion Criteria:

* Unable to give consent
* Crohn's disease
* Does not meet inclusion criteria
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Urine for PGEm Levels | Day of colonoscopy procedure

SECONDARY OUTCOMES:
Blood for CRP | Day 1
Stool for fecal calprotectin | At least 2 days before colonoscopy procedure (prior to bowel prep)
MAYO disease activity score | Day of colonoscopy procedure
Routine colonoscopy for assessment of disease activity | 1-3 weeks after consent

CONTACTS AND LOCATIONS:
Overall Officials: David A. Schwartz, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States